CLINICAL TRIAL: NCT03837977
Title: A Multi-centre, Randomised, Parallel Group, Open-label, Phase II, Single-stage Selection Trial of Liposomal Irinotecan (Nal-IRI) and 5-fluorouracil (5-FU)/Folinic Acid or Docetaxel as Second-line Therapy in Patients With Progressive Poorly Differentiated Extra-pulmonary Neuroendocrine Carcinoma (NEC))
Brief Title: Second-line Therapy for Patients With Progressive Poorly Differentiated Extra-pulmonary Neuroendocrine Carcinoma
Acronym: NET02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Leeds (Other); Servier (Industry); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp116
Record Dates: First submitted 2018-09-27; First posted 2019-02-12 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Oncology; Neuroendocrine Carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Neuroendocrine | interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin; Docetaxel

STUDY DESIGN:
Intervention Model Description: The study is a randomised controlled trial. One hundred and two eligible participants will be randomised (1:1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nal-IRI, 5-FU and racemic folinic acid (Active Comparator): liposomal Irinotecan (naI-IRI) (80mg/m*2 intravenously over 90 minutes (± 10 minutes) prior to Fluorouracil (5-FU) 5-FU 2400 mg /m*2 BSA infusor over 46 hours racemic folinic acid (as per local standard practice) every 14 days
  Interventions: Drug: Liposomal Irinotecan; Drug: Fluorouracil; Drug: Folinic Acid
- docetaxel (Active Comparator): 75mg/m*2 intravenously over 60 minutes) every 21 days]
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Liposomal Irinotecan — Arm I
  Other Names: Onivyde
  Arms: nal-IRI, 5-FU and racemic folinic acid
Drug: Fluorouracil — Arm I
  Arms: nal-IRI, 5-FU and racemic folinic acid
Drug: Folinic Acid — Arm I
  Arms: nal-IRI, 5-FU and racemic folinic acid
Drug: Docetaxel — Arm II
  Arms: docetaxel

SUMMARY:
There is currently no standard treatment beyond first-line etoposide/platinum-based chemotherapy in patients with progressive poorly differentiated extra-pulmonary neuroendocrine carcinoma. Therefore the treatment of patients whose disease progresses on or after this first-line treatment is an area of unmet need.

Combination regimens such as irinotecan/5-fluorouracil/folinic acid are a second-line treatment option currently used in Europe and world-wide for this subset of patients. However, there is currently no trial evidence supporting this treatment regimen in these patients.

Results of the NAPOLI-1 phase III trial of liposomal irinotecan in the treatment of patients with metastatic pancreatic adenocarcinoma after gemcitabine-based therapy reported improved survival for those patients who received a combination of liposomal irinotecan with 5-FU/folinic acid compared to those patients who received 5-FU/folinic acid alone. Liposomal irinotecan has been found to show an improved distribution into tumour tissue in comparison to irinotecan, and this may have clinical benefit in patients with extra-pulmonary neuroendocrine carcinoma.

Docetaxel is standardly used as a second-line treatment option in patients with small cell lung cancer who have progressed on primary etoposide-platinum combination therapy. Therefore this drug could also have clinical benefit in patients with extra-pulmonary neuroendocrine carcinoma as the biology of the disease is similar to small cell lung cancer.

The overall aim of the NET-02 trial is to select a treatment for continuation to a Phase III trial. The intention of the trial is to determine whether liposomal irinotecan/5-fluorouracil/folinic acid and docetaxel are sufficiently active in this population of patients. If both treatments are found to be efficacious, selection criteria will be applied to select a treatment to take forward.

102 eligible participants will be randomised to receive either liposomal irinotecan/5-fluorouracil/folinic acid given every 14 days, or docetaxel given every 21 days. Participants will be treated for a minimum of 6 months or until discontinuation of treatment as per protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and life expectancy ≥3 months.
2. Diagnosed with poorly differentiated (as defined by the World Health Organisation in 2010, Ki 67 ≥20%) extra-pulmonary neuroendocrine carcinoma (NEC grade 3, confirmed by histology). (Carcinoma of unknown primary is allowed if lung primary has been excluded following review by the multi-disciplinary team).
3. Prior treatment with first-line platinum-based chemotherapy for NEC in the advanced setting and ≥28 days from Day 1 of the previous treatment cycle.
4. Documented radiological evidence of disease progression OR discontinuation of first-line platinum-based chemotherapy due to intolerance.
5. Measurable disease according to RECIST 1.1
6. Eastern Co-operative Oncology Group (ECOG) performance status ≤2
7. Adequate renal function with serum creatinine ≤1.5 times upper limit of normal (ULN) and creatinine clearance ≥50ml30ml/min according to Cockroft-Gault or Wright formula. If the calculated creatinine clearance is less than 30 ml/min, glomerular filtration rate (GFR) may be assessed using either Cr51-EDTA or 99mTc-DTPA clearance method to confirm if GFR is ≥30 ml/min).
8. Adequate haematological function: Hb ≥90g/L, WBC ≥3.0 x 109/L, ANC ≥1.5 x 109/L, platelet count ≥100 x 109/L.
9. Adequate liver function: serum total bilirubin 1.5 x ULN (biliary drainage is allowed for biliary obstruction) and ALT and/or AST 2.5 x ULN in the absence of liver metastases, or 5 x ULN in the presence of liver metastases.
10. A negative pregnancy test is required at registration in women of childbearing potential.
11. Men and women of reproductive potential must agree to use a highly effective form of contraception during the study and for 6 months following the last dose of trial treatment. In addition, male participants should use a condom during study participation and for 6 months following the last dose of trial treatment.
12. Patients must be able to provide written informed consent.
13. Patients must be able and willing to comply with the terms of the protocol.

Exclusion Criteria:

1. Known or suspected allergy or hypersensitivity reaction to any of the components of study treatment or their excipients.
2. Use (including self-medication) within one week of randomisation and for the duration of the study of any of the following: St. John's wort, grapefruit, Seville oranges, medicines known to inhibit UGT1A1 (e.g. atazanavir, gemfibrozil, indinavir) and medicines known to inhibit or induce either CYP3A4 or CYP3A5
3. Previous treatment (for neuroendocrine carcinoma) with any of the components of combination chemotherapy regimens detailed in this study (nal-IRI or 5-FU or irinotecan or topoisomerase inhibitors or taxane-based therapy).
4. Incomplete recovery from previous therapy in the opinion of the investigator (surgery/adjuvant therapy/radiotherapy/chemotherapy in advanced setting), including ongoing peripheral neuropathy of Common Terminology Criteria for Adverse Events (CTCAE) grade 2 from previous platinum-based therapy.
5. Concurrent palliative radiotherapy involving target lesions used for this study (<28 days from discontinuation of radiotherapy). Radiotherapy for non-target lesions is allowed if other target lesions are available outside the involved field.
6. Patients must not have a history of other malignant diseases (within the previous 3 years, and there must be no evidence of recurrence), other than:

   * Extra-pulmonary neuroendocrine carcinoma.
   * Non-melanoma skin cancer where treatment consisted of resection only or radiotherapy.
   * Ductal carcinoma in situ (DCIS) where treatment consisted of resection only.
   * Cervical carcinoma in situ where treatment consisted of resection only.
   * Superficial bladder carcinoma where treatment consisted of resection only.
7. Documented brain metastases, unless adequately treated (surgery or radiotherapy only), with no evidence of progression and neurologically stable off anticonvulsants and steroids.
8. Clinically significant gastrointestinal disorder (in the opinion of the treating clinician) including hepatic disorders, bleeding, inflammation, obstruction, or diarrhoea ≥CTCAE grade 1 (at time of study entry).
9. Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) less than 6 months before inclusion.
10. New York Heart Association (NYHA) Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure .
11. Severe bone marrow failure or bone marrow depression after radiotherapy or treatment with other antineoplastic agents (defined as haematological values of haemoglobin or white blood cells or neutrophils or platelets not meeting inclusion criteria).
12. Known active hepatitis B virus, hepatitis C virus or HIV infection.
13. Active chronic inflammatory bowel disease.
14. Breastfeeding women.
15. Evidence of severe or uncontrolled systemic diseases which, in the view of the treating clinician, makes it undesirable for the patient to participate in the trial.
16. Evidence of significant clinical disorder or laboratory finding which, in the opinion of the treating clinician, makes it undesirable for the patient to participate in the trial.
17. Medical or psychiatric conditions that impair the ability to give informed consent.
18. Any other serious uncontrolled medical conditions (in the opinion of the treating clinician).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Progression-free survival defined as a binary outcome (progression-free or not) | treatment start date until 6 months, assessed at 8 weekly intervals by CT scan

SECONDARY OUTCOMES:
Progression-free survival defined as time from randomisation to progression or death from any cause. | randomisation until 6 months after the last participant is randomised (end of trial), assessed at 8 weekly intervals by CT scan and death is continuously assessed
  Individuals will be censored if they are lost to follow-up or still alive and progression-free at the time of analysis.
Overall survival defined as time from randomisation to death from any cause. | randomisation until 6 months after the last participant is randomised (end of trial), death is continuously assessed
  Individuals will be censored if they are lost to follow-up or still alive and progression-free at the time of analysis.
Objective response rate defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. | start of treatment until 6 months after the last participant is randomised (end of trial)
Toxicity defined as the number of participants with treatment-related adverse events as assessed by common terminology criteria for adverse events (CTCAE) v5.0. | treatment start date until 6 months after the last participant is randomised (end of trial), assessed at 2 (nal-IRI/5-FU/folinic acid) or 3 (docetaxel) weekly intervals
Quality of life assessed according to the patient reported outcome measures; European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 | randomisation until 6 months after the last participant is randomised (end of trial), assessed at 6 weekly intervals
Neuron-specific enolase (NSE) measurements. | baseline until 6 months after the last participant is randomised (end of trial), assessed at 6 weekly intervals
Quality of life assessed according to the patient reported outcome measures; European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) GINET21. | randomisation until 6 months after the last participant is randomised (end of trial), assessed at 6 weekly intervals

CONTACTS AND LOCATIONS:
Overall Officials: Mairead McNamara, Principal Investigator — The Christie NHS Foundation Trust, The University of Manchester
Locations (4):
- United Kingdom (4):
  - The Beaston West of Scotland Cancer Center, NHS Greater Glasgow and Clyde, Glasgow
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Weston Park Hospital, Sheffield Teaching Hospitals, NHS Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data datasets generated and/or analysed during the current study will be available upon request from the Clinical Trials Research Unit, University of Leeds (contact CTRU-DataAccess@leeds.ac.uk in the first instance).
  No individual participant data will be released before an appropriate agreement is in place setting out the conditions of release. The agreement will govern data retention, usually stipulating that data recipients must delete their copy of the released data at the end of the planned project.
  The CTRU encourages a collaborative approach to data sharing, and believe it is best practice for researchers who generated datasets to be involved in subsequent uses of those datasets. Recipients of trial data for secondary research will also receive data dictionaries, copies of key trial documents and any other information required to understand and reuse the released datasets.
Time Frame: Data will be made available at the end of the trial, i.e. usually when all primary and secondary endpoints have been met and all key analyses are complete. Data will remain available from then on for as long as CTRU retains the data.
Access Criteria: CTRU makes data available by a 'controlled access' approach. Data will only be released for legitimate secondary research purposes, where the Chief Investigator, Sponsor and CTRU agree that the proposed use has scientific value and will be carried out to a high standard (in terms of scientific rigour and information governance and security), and that there are resources available to satisfy the request. Data will only be released in line with participants' consent, all applicable laws relating to data protection and confidentiality, and any contractual obligations to which the CTRU is subject. The conditions of release for aggregate data may differ from those applying to individual participant data. Requests for aggregate data should also be sent to the above email address to discuss and agree suitable requirements for release.

REFERENCES:
- [Derived] McNamara MG, Swain J, Craig Z, Sharma R, Faluyi O, Wadsley J, Morgan C, Wall LR, Chau I, Reed N, Sarker D, Margetts J, Krell D, Cave J, Sothi S, Anthoney A, Bell C, Patel A, Oughton JB, Cairns DA, Mansoor W, Lamarca A, Hubner RA, Valle JW. NET-02: a randomised, non-comparative, phase II trial of nal-IRI/5-FU or docetaxel as second-line therapy in patients with progressive poorly differentiated extra-pulmonary neuroendocrine carcinoma. EClinicalMedicine. 2023 Jun 2;60:102015. doi: 10.1016/j.eclinm.2023.102015. eCollection 2023 Jun. PMID 37287870
- [Derived] Craig Z, Swain J, Batman E, Wadsley J, Reed N, Faluyi O, Cave J, Sharma R, Chau I, Wall L, Lamarca A, Hubner R, Mansoor W, Sarker D, Meyer T, Cairns DA, Howard H, Valle JW, McNamara MG. NET-02 trial protocol: a multicentre, randomised, parallel group, open-label, phase II, single-stage selection trial of liposomal irinotecan (nal-IRI) and 5-fluorouracil (5-FU)/folinic acid or docetaxel as second-line therapy in patients with progressive poorly differentiated extrapulmonary neuroendocrine carcinoma (NEC). BMJ Open. 2020 Feb 5;10(2):e034527. doi: 10.1136/bmjopen-2019-034527. PMID 32029495